CLINICAL TRIAL: NCT04347278
Title: Observational Study of Follow-up of Hospitalized Patients Diagnosed With COVID-19 to Evaluate the Effectiveness of the Drug Treatment Used to Treat This Disease. COVID-19 Registry
Acronym: RegCOVID19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Instituto de Investigación Marqués de Valdecilla (Other)
Collaborators: Hospital Universitario Marqués de Valdecilla (Other); Hospital Universitario de Canarias (Other); Hospital San Pedro de Alcantara (Other)
Responsible Party: Sponsor
Other Study IDs: IDI-REM-2020-1
Record Dates: First submitted 2020-04-03; First posted 2020-04-15 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: SARS-CoV-2
Keywords: COVID19; ICU
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients receiving treatment for COVID19
  Interventions: Drug: Patients with the treatment agains COVID19

INTERVENTIONS:
Drug: Patients with the treatment agains COVID19 — Data will be collected from patients who receive any of the treatments included in the "Technical Document. Manejo clínico del COVID-19: tratamiento médico" of the Ministry of Health, and "Tratamientos disponibles para el manejo de la infección respiratoria por SARS-CoV-2" of the AEMPS, either as antivirals or as treatment of the inflammatory process in patients with SARS, or others as they arise.

SUMMARY:
The infection caused by COVID19 worldwide makes it necessary to monitor drugs administered for the treatment of patients hospitalized with SARS-CoV-2. In order to know more about the efficacy and safety of the treatments used, researchers from the Cantabrian health service have developed an observational study, in the form of an ambispective registry, in which clinical data from patients treated with the different drugs currently recommended by the Spanish Agency of Medicines and Health Products (SAMHP) and the Ministry of Health, or others that may arise, are collected and analyzed.

Although the conduct of clinical trials is a priority at this time, we cannot lose the clinical experience that is currently being generated, which may allow us to improve the therapeutic strategies for future patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients of any age and gender, including minors and pregnant women.
* Hospital admission with diagnosis of COVID-19 according to clinical and microbiological criteria established by the Health Authorities and clinical practice (these may be modified based on the "Technical Document. Clinical management of COVID-19: hospital care" of the Ministry of Health).
* Patients receiving any specific treatment for COVID-19 disease (according to the "Technical Document. Clinical management of COVID-19: medical treatment" of the Ministry of Health, and "Available treatments for the management of respiratory infection by SARS-CoV-2" of the AEMPS).
* Patients admitted but not receiving specific treatment for COVID-19 disease

Exclusion Criteria:

* Patients who do not wish to give informed consent once requested.

Ages: 1 Year to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The subject of the study is any person diagnosed with COVID-19 who is admitted to a hospital either as an inpatient or in an intensive care unit (ICU).
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-04-22 (Actual); Primary Completion 2021-10-15 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of current drug treatments for hospitalized patients with SARS-CoV-2 infection (COVID-19 patients) in routine clinical practice | 6 months
  Measured in terms of clinical recovery

SECONDARY OUTCOMES:
Risk factors or modifiers of pharmacological effect such as demographic characteristics, comorbidity or underlying pathology, concomitant medication. | 6 months
Information on the patterns of use of these drugs (dose, duration of treatment, | 6 months
  to know the use according to the Ministry of Health Technical Document
Adverse events | 6 months
  Adverse effects of the medicines used
Time of hospital admission and/or stay in ICU and maximum severity reached. | 6 months
Treatments for SARS-CoV-2 positive patients not described in the protocol | 6 months
  Determine the evolution of the treatments
healthy survey for patients after their recovery/discharge from hospital. | 6 months
  It is composed of 10 items, with scores from 0 (worst health) to 100 points (best health)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Marqués de Valdecilla, Santander, Cantabria, Spain

IPD SHARING:
Plan to Share IPD: No